CLINICAL TRIAL: NCT04312451
Title: Prospective Cohort of Patients With Critical Limb Ischemia Undergoing Revascularization
Acronym: CLI ENDOVASC
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CLI ENDOVASC
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripheral Arterial Occlusive Disease is associated with a high risk of cardiovascular events. The critical ischemia stage represents the most severe stage of Peripheral Arterial Occlusive Disease, associated with decubitus pain and / or foot ulceration. The severity of this arterial involvement involves functional prognosis of the lower limb with a high risk of amputation, and the vital prognosis of the patient. In these patients, the rate of amputation and mortality at 1 year can reach 20%. Therefore, the goal of management in a multidisciplinary setting is limb salvage and improvement of the patient's vital prognosis.

In the vascular medicine department, the indication and modalities of the revascularization procedure are discussed in a multidisciplinary consultation meeting. Surgical revascularization by distal bypass requires venous material that can be used, a receiving artery without diffuse lesions, in direct continuity with the arterial network of the foot, and the absence of co-morbidities against general anesthesia. With the modernization and development of endovascular equipment dedicated to the hamstrings, the interventional radiology techniques in the management of critical ischemia allow the treatment of one or more arterial axes as well as a very distal revascularization in the arteries. of the foot with less morbidity-mortality compared to surgery, especially in patients the most fragile patients. Since 2013, the endovascular revascularization procedures performed by the interventional radiology team have been an integral part of the management of patients with peripheral arterial disease of the lower limbs monitored in the vascular medicine department. The hospital is therefore a privileged place to observe the long-term impact of this medical care on the future of patients with different stages of severity of arterial disease.

The objective of this prospective study is to assess the vital prognosis, limb salvage and associated prognostic factors in patients with critical ischemia supported by endovascular revascularization in the vascular medicine service of the GHPSJ. The objective of this cohort study is to build a database on critical ischemia in hospitalized patients, to judge the management, monitoring and prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Man or Woman whose age is ≥ 18 years old
* Patient with critical lower limb ischemia defined by the existence of decubitus pain or a wound (foot ulcer or gangrene) evolving for more than 2 weeks associated with hemodynamic criteria (systolic toe pressure <30 mm Hg and / or systolic ankle pressure <50 mm Hg).
* Hospitalized in the vascular medicine department
* Endovascular revascularization gesture discussed and confirmed by multidisciplinary staff

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patients objecting to the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are hospitalized in the vascular medicine department of the Paris Saint-Joseph Hospital Group, for the management of critical ischemia of the lower limbs with decision to revascularize by endovascular route for leg rescue, after discussion in multidisciplinary staff (associating vascular physicians, vascular surgeons and interventional radiologists).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
Survival rate without major amputation | Year 1
  This outcome measure the survival rate without major amputation at 1 year.

SECONDARY OUTCOMES:
Prevalence of intraoperative deaths | Day 1
  This outcome measures the prevalence of intraoperative deaths.
Prevalence of intraoperative cardiovascular events | Day 1
  This outcome measures the prevalence of intraoperative cardiovascular events.
Prevalence of intraoperative deaths, at 1 year | Year 1
  This outcome measures the prevalence of intraoperative deaths, at 1 year after the surgery.
Prevalence of intraoperative cardiovascular events, at 1 year | Year 1
  This outcome measures the prevalence of intraoperative cardiovascular events at 1 year after the surgery.
Healing rate | Year 1
  This outcome measures the healing rate, 1 year after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra YANNOUTSOS, mD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Savji N, Rockman CB, Skolnick AH, Guo Y, Adelman MA, Riles T, Berger JS. Association between advanced age and vascular disease in different arterial territories: a population database of over 3.6 million subjects. J Am Coll Cardiol. 2013 Apr 23;61(16):1736-43. doi: 10.1016/j.jacc.2013.01.054. Epub 2013 Apr 2. PMID 23500290
- [Result] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Result] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Result] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I, Document Reviewers, Widimsky P, Kolh P, Agewall S, Bueno H, Coca A, De Borst GJ, Delgado V, Dick F, Erol C, Ferrini M, Kakkos S, Katus HA, Knuuti J, Lindholt J, Mattle H, Pieniazek P, Piepoli MF, Scheinert D, Sievert H, Simpson I, Sulzenko J, Tamargo J, Tokgozoglu L, Torbicki A, Tsakountakis N, Tunon J, Vega de Ceniga M, Windecker S, Zamorano JL. Editor's Choice - 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Mar;55(3):305-368. doi: 10.1016/j.ejvs.2017.07.018. Epub 2017 Aug 26. No abstract available. PMID 28851596
- [Result] Romiti M, Albers M, Brochado-Neto FC, Durazzo AE, Pereira CA, De Luccia N. Meta-analysis of infrapopliteal angioplasty for chronic critical limb ischemia. J Vasc Surg. 2008 May;47(5):975-981. doi: 10.1016/j.jvs.2008.01.005. Epub 2008 Apr 18. PMID 18372148
- [Result] Salas CA, Adam DJ, Papavassiliou VG, London NJ. Percutaneous transluminal angioplasty for critical limb ischaemia in octogenarians and nonagenarians. Eur J Vasc Endovasc Surg. 2004 Aug;28(2):142-5. doi: 10.1016/j.ejvs.2004.03.023. PMID 15234694
- [Result] Faglia E, Mantero M, Caminiti M, Caravaggi C, De Giglio R, Pritelli C, Clerici G, Fratino P, De Cata P, Dalla Paola L, Mariani G, Poli M, Settembrini PG, Sciangula L, Morabito A, Graziani L. Extensive use of peripheral angioplasty, particularly infrapopliteal, in the treatment of ischaemic diabetic foot ulcers: clinical results of a multicentric study of 221 consecutive diabetic subjects. J Intern Med. 2002 Sep;252(3):225-32. doi: 10.1046/j.1365-2796.2002.01015.x. PMID 12270002